CLINICAL TRIAL: NCT02913118
Title: Adjunctive Therapy of Andrographolid Sulfonatein Community Acquired Pneumonia: A Multicenter Randomized Controlled Clinical Trial
Brief Title: Adjunctive Therapy of Andrographolid Sulfonatein Community Acquired Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingfeng Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: QF-CAP-20160402
Record Dates: First submitted 2016-09-12; First posted 2016-09-23 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Cephalosporins; Azithromycin; Minocycline; Doxycycline; Fluoroquinolones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard antibiotic treatment +AS injection (Experimental): Andrographolid Sulfonate Injection (AS Injection) plus one of 3 antibiotics in China CAP Guideline
  Interventions: Drug: Andrographolid Sulfonate Injection (AS Injection); Drug: Cephalosporin; Drug: Azithromycin, Minocycline or Doxycycline; Drug: Amoxicillin-clavulantic acid; Drug: Fluoroquinolones
- standard antibiotic treatment + AS placebo (Placebo Comparator): AS placebo (NS injection) plus one of 3 antibiotics in China CAP Guideline
  Interventions: Drug: Cephalosporin; Drug: Azithromycin, Minocycline or Doxycycline; Drug: Amoxicillin-clavulantic acid; Drug: Fluoroquinolones; Drug: Placebo

INTERVENTIONS:
Drug: Andrographolid Sulfonate Injection (AS Injection)
  Arms: standard antibiotic treatment +AS injection
Drug: Cephalosporin
Drug: Azithromycin, Minocycline or Doxycycline
Drug: Amoxicillin-clavulantic acid
Drug: Fluoroquinolones
Drug: Placebo
  Arms: standard antibiotic treatment + AS placebo

SUMMARY:
Adjunctive Therapy of AndrographolidSulfonate in Community Acquired Pneumonia: A Multicenter, Randomized,Double-blinded, Placebo Controlled Clinical Trial. The hypothesis is that combination therapy with Andrographolid Sulfonatein injection and antibacterial is significantly better than antibacterial alone in achieving clinical stability among hospitalized CAP patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75 years, no gender restrictions.
* Voluntary participation, all participants provide written informed consent.
* Volunteers are hospitalized patients
* Patients are hospitalized for community acquired pneumonia with T≥38°C within 24 hours before being enrolled Diagnosis of CAP(Chinese Guideline for Diagnosis and Management of Community Acquired Pneumonia in Adults 2016)

  1. Pneumonia that is acquired in community
  2. Symptoms and signs of pneumonia:

  <!-- -->

  1. Presence of cough, expectoration or exacerbation of chronic airways disease, with or without purulent sputum/chest pain/dyspnea/hemoptysis.
  2. Presence offever.
  3. Lung consolidation and/or moist rales.
  4. Peripheral blood（WBC）>10×109/L or <4×109/L, with or without nuclear left shift; 3. Chest radiograph shows new ground-glass opacity, patchy infiltration, consolidation or interstitial changes, with or without pleural effusion.

Patients who meet 1,3 and any one item in 2, exclude one of the following are clinically classified as CAP: pulmonary tuberculosis, cancer, non-infectious interstitial lung disease, pulmonary edema, atelectasis, pulmonary embolism, pulmonary eosinophilia and pulmonary vasculitis.

* CURB 65≥1 point,Each risk factor scores one point, for a maximum score of 5:

  * Confusion of new onset
  * Blood Urea nitrogen greater than 7 mmol/l (19 mg/dL)
  * Respiratory rate of 30 breaths per minute or greater
  * Blood pressure less than 90 mmHg systolic or diastolic blood pressure 60 mmHg or less
  * Age 65 or older
* Within 72 hours after symptom onset

Exclusion Criteria:

* Known allergy to AS
* Pregnant or breast-feeding
* Heart dysfunction, NYHA III-IV class
* Hematological system diseases, such as lymphoma, leukemia, agranulocytosis (neutrophil count< 0.5×109/L).
* Autoimmune diseases and disease active
* Terminal malignant tumor
* Long-term treatment of high dose corticosteroids (prednisone 10mg/d ≥2 weeks) or immunosuppressive agents
* Inflammatory bowel disease, such as Crohn's disease, ulcerative colitis
* Chronic renal failure, eGFR<50 ml/min/1.73m2
* Severe liver function damage, ALT or AST greater than or equal to 2 times the upper limit of normal
* Hypernatremia, serum sodium≥145mmol/L
* Diagnosis as severe pneumonia:

Diagnostic criteria of severe pneumonia: patients who meet one major criteria or at least 3 of these minor criteria are classified as severe cases: Major criteria:①the need for invasive mechanical ventilation②sepsis shock after active fluid resuscitation still need vasoactive drugs; Minor criteria:①respiratory rate >30 breaths/min, ②PaO2/FiO2≤250mmHg（1mmHg=0.133kPa）, ③multilobar infiltrates, ④confusion or/andunorientation, ⑤bloodurea nitrogen level≥20mg/dl（7.14mmol/L）, ⑥systolic pressure <90mmHg need active fluid resuscitation

* Defervescence by using corticosteroid after symptom onset.
* Patients who participated another intervention study within a month
* Other conditions not suitable for inclusion according to the investigator' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
time to clinical stability | 14 days
number of study participants with treatment-related adverse events as assessed by CTCAE v4.0 | 14 days
  symptoms and signs, blood and urine routine, liver and kidney function monitoring, ECG, side effects of long-time using of antibiotics

SECONDARY OUTCOMES:
the duration of fever | 14 days
the initial treatment failure rate | 14 days
length of stay in hospital | 14 days
questionnaire for hospitalization expenses | 14 days
the duration of intravenous antibiotic treatment | 14 days
the rate of diarrhea and intestinal dysbacteriosis | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Professor, Principal Investigator — China-Japan Friendship Hospital; Bin Cao, Professor, Principal Investigator — China-Japan Friendship Hospital; Jin Chen, Professor, Principal Investigator — Fu Xing Hospital, Capital Medical University; Yuguang Wang, Professor, Principal Investigator — Beijing Hospital of TCM; Li Gu, Professor, Principal Investigator — Beijing Chao Yang Hospital; Zhenyang Xu, Professor, Principal Investigator — Capital Medical University; Yan Yi, Professor, Principal Investigator — First Hospital of China Medical University; Wei Zhang, Professor, Principal Investigator — The First Affiliated Hospital of Nanchang University; Shufeng Xu, Professor, Principal Investigator — First Hospital of Qinhuangdao; Bo Liu, Professor, Principal Investigator — The Central Hospital of ZiBo City; Jie Cao, Professor, Principal Investigator — Tianjin Medical University General Hospital; Yuping Li, Professor, Principal Investigator — The First Affiliated Hospital of Wenzhou University; Xuedong Liu, Professor, Principal Investigator — Qingdao Municipal Hospital; Hong Fan, Professor, Principal Investigator — West China Hospital; Zhigang Cai, Professor, Principal Investigator — The Second Hospital of Hebei Medical University; Xinri Zhang, Professor, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Xin Su, Professor, Principal Investigator — Nanjing General Hospital
Locations (16):
- China (16):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Hospital of TCM, Beijing, Beijing Municipality
  - Beijing LuHe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fu Xing Hospital, Capital Medical Unviersity, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Wenzhou University, Wenzhou, Fujian
  - First Hospital of QinHuangDao, Qinhuangdao, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanjing General Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The Central Hospital of ZiBo City, Zibo, Shandong
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Shang LH, Fan GH, Chen LP, Liu JH, Wang XG, Liu B, Tian GZ, Chen XS, Yu JX, Yang GR, Su X, Liu XD, Li YP, Xu SF, Lin YH, Cao J, Zhang W, Feng WS, Cai ZG, Wang QH, Wang JX, Wang YG, Chen J, Zhang YX, Cui XJ. Andrographolide Sulfonate Injection for Adjunctive Treatment of Non-severe Community-Acquired Pneumonia in Adults: A Multicenter, Double-Blind, Randomized Controlled Trial. Chin J Integr Med. 2026 Jan 5. doi: 10.1007/s11655-025-3932-8. Online ahead of print. PMID 41489779